CLINICAL TRIAL: NCT05852327
Title: Risk Stratifying COPD Exacerbations: a Prospective Study
Brief Title: Risk Stratifying COPD Exacerbations
Acronym: ProECOPD_23
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Wong Charles, Associate Consultant, Department of Medicine, Pamela Youde Nethersole Eastern Hospital
Other Study IDs: ProECOPD_23
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD: Subjects with COPD exacerbation
  Interventions: Other: Observation only

INTERVENTIONS:
Other: Observation only — Observation only

SUMMARY:
To identify clinical characteristics on presentation which predict differential outcomes in patients with exacerbation of COPD.

DETAILED DESCRIPTION:
Exacerbations of COPD (ECOPD) are heterogenous but are often considered as a single clinical entity. Clinical characteristics on presentation may predict outcome of patients with ECOPD.

DECAF score was previously proposed to predict in-hospital mortality but has not been validated in Asian subjects. ROME classification was recently proposed to better risk stratify ECOPD according to symptoms, physiological parameters and laboratory findings on admission, but no prospective validation study is available so far.

This study aims to identify clinical characteristics on presentation to predict outcome of patients with ECOPD.

ELIGIBILITY:
Inclusion Criteria:

* Background history of COPD, defined by the GOLD 2023 guidelines
* Presented with exacerbation of COPD, defined by the GOLD 2023 guidelines
* Age >= 18 years old
* Informed consent available

Exclusion Criteria:

* Age < 18 years old
* No informed consent

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 500 subjects with COPD exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 3-month
  Number of patients died during hospitalization of ECOPD
3-month mortality | 3-month
  Number of patients died 3 months after ECOPD
Recurrent ECOPD | 3-month
  Number of patients with recurrent ECOPD post-discharge
Viral etiology | 3-month
  Frequency of various viral etiology identified during ECOPD
Bacterial etiology | 3-month
  Frequency of various bacterial etiology identified during ECOPD

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Charles Wong, Hong Kong, Other
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No